CLINICAL TRIAL: NCT05568862
Title: The Characteristics of Ureteric Jet Doppler Waveforms and Factors Affecting Them in Patients With Spinal Cord Injury
Brief Title: Ureteric Jet Doppler Waveforms in Patients With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: ik
Record Dates: First submitted 2022-10-01; First posted 2022-10-06 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spinal cord injury: patient with spinal cord injury
  Interventions: Diagnostic Test: Doppler ultrasound, Urodynamic assessment.; Diagnostic Test: Urodynamic assessment.
- no spinal cord injury: patient without spinal cord injury
  Interventions: Diagnostic Test: Doppler ultrasound, Urodynamic assessment.

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound, Urodynamic assessment. — The patients included in the study group were given 600 cc of water in the morning and the Doppler ultrasound was performed 30 minutes later
Diagnostic Test: Urodynamic assessment. — A transurethral double lumen catheter was used to measure intravesical pressure in the urodynamic unit for the patients in the study group immediately after the use of the Doppler USG
  Groups: spinal cord injury

SUMMARY:
Urinary dysfunction is very common in individuals with spinal cord injury. The urine flowing from the collecting ducts to the renal calyx stretches the calyces. ANS controlled peristaltic contractions originate in the proximal renal pelvis and travel down the ureters, pushing urine from the renal pelvis towards the bladder. The urine bolus delivered from the kidneys through the peristaltic contraction of the ureter creates an image called ureteric jet. Using the Doppler analysis of ureteral jets, previous studies have examined the changes in the ureteric jet pattern in pathological conditions such as the diagnosis of normal ureteral physiology.

DETAILED DESCRIPTION:
This cross-sectional study was conducted at a tertiary rehabilitation center. Eighteen spinal cord injury patients who met the inclusion criteria and 24 healthy volunteers were included in the study. The appearance of üreteric jet form and bladder wall thicknesses were obtained by urinary Doppler ultrasound both in patient and control groups. Detrusor pressure and bladder volume were measured only in patient group during urodynamic assessment.

ELIGIBILITY:
The case group

Inclusion Criteria:

* With signs of upper motor neuron lesion,
* Suprasacral spinal cord injury,
* Normal urinary ultrasound findings
* Planned urodynamics

Exclusion Criteria:

* Neurological disease other than spinal cord injury
* Urinary tract infection
* Urinary obstruction
* History of urinary tract Stones
* Diabetes, hypertension
* History of urinary surgery,
* Sacral injury
* Second motor neuron lesions (such as cauda equina, or cauda conus)

The control group

Inclusion Criteria:

• Normal urinary ultrasonography

Exclusion Criteria:

* Neurological disease
* Urinary tract infection
* Urinary obstruction
* History of urinary tract Stones
* Diabetes, hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal cord injury patients who were hospitalized in the spinal cord injury Rehabilitation Unit of our rehabilitation center and 32 no spinal cord injury who presented at outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
doppler USG | 15-30 minute
  The patients included in the study group were given 600 cc of water in the morning and the Doppler USG was performed 30 minutes later
Urodynamic assessment. | 30 minute
  A transurethral double lumen catheter was used to measure intravesical pressure in the urodynamic unit

CONTACTS AND LOCATIONS:
Overall Officials: İlkay Karabay, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler PMR, Training and Research Hospital, Department of PMR, Ankara, Çankaya, Turkey (Türkiye)